CLINICAL TRIAL: NCT03846089
Title: A Propensity Score Matched Pair Analysis of Retrograde Reperfusion Versus Antegrade Liver Transplant Reperfusion
Brief Title: Retrograde Reperfusion Versus Antegrade Liver Transplant Reperfusion
Status: Withdrawn | Type: Observational
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Vivian McAlister, Professor of Surgery, London Health Sciences Centre
Other Study IDs: 106793
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Liver Transplant Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrograde reperfusion: After completion of the inferior vena cava anastomosis, the clamps were removed to allow retrograde reperfusion of the graft.
  Interventions: Procedure: Graft reperfusion
- Antegrade reperfusion: After completion of the inferior vena cava anastomosis, the portal vein anastomosis is completed and then the clamps were removed to allow antegrade reperfusion of the graft.
  Interventions: Procedure: Graft reperfusion

INTERVENTIONS:
Procedure: Graft reperfusion — antegrade (forward) or retrograde (backward) blood reperfusion of the liver graft

SUMMARY:
A retrospective cohort analysis was performed comparing patients that had intra operative antegrade liver reperfusions versus patients that had retrograde liver perfusion.

DETAILED DESCRIPTION:
A retrospective cohort analysis was performed comparing patients that had intra operative antegrade liver reperfusions versus patients that had retrograde liver perfusion. Antegrade Reperfusion(ATR) group: after completing the caval replacement or piggy-back, for IVC anastomosis, Portal vein (PV) anastomosis was done with a running suture as normal fashion, then it was followed by the removal the clamps, starting by the supra hepatic VC, followed by the PV clamp and finally the infrahepatic VC. It was followed by arterial anastomosis and the biliary anastomosis (duct-to-duct if possible). Retrograde group (RETR): after completing the piggyback the IVC was declamped immediately and retrograde low pressure reperfusion of the graft with low oxygenated venous blood was established. Central venous pressure was intended to be higher than in 8 mmHg to enable appropriate retrograde reperfusion in the transplanted liver. Significant venous backflow via portal vein appears immediately after declamping. Venous bleeding from the liver except portal backflow was stopped immediately after declamping the venous anastomosis, as appropriate. Portal vein anastomosis was performed using running suture. It was followed by arterial anastomosis and the biliary anastomosis (duct-to-duct if possible). The endpoints are patient survival and graft survival at 1, 3,5, 10 years post liver transplantation in both groups. To adjust for a selection bias, we will perform a propensity score analysis.

ELIGIBILITY:
Inclusion Criteria:

* all liver transplantations between 1 Jan 2002 and 31 Dec 2005

Exclusion Criteria:

* liver retransplantation
* multiorgan transplantation
* ABO incompatible transplantation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have undergone transplantation of the liver at LHSC.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Graft survival | From date of transplantation until the date of next transplantation or date of death from any cause, whichever came first, assessed up to 300 months
  Average length of time the liver graft remains in a living recipient regardless of function

SECONDARY OUTCOMES:
Patient survival | From date of transplantation until the date of death from any cause assessed up to 300 months
  Average length of time a recipient is alive regardless of presence of the second liver

CONTACTS AND LOCATIONS:
Overall Officials: Vivian McAlister, Principal Investigator — London Health Sciences Center

IPD SHARING:
Plan to Share IPD: Yes
Study mechanisms and de-identified subject level data will be shared with researchers who contact the principal investigator.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: From the time of publication for 5 years
Access Criteria: By contacting the PI and with permission of the REB